CLINICAL TRIAL: NCT03908086
Title: Incidence and Risk Factors of Staphylococcus Aureus Bacteremia in Patients With Rheumatoid Arthritis Compared With the General Population
Brief Title: Bloodstream Infections in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Sabine Dieperink (Other)
Collaborators: University of Copenhagen (Other); University of Aarhus (Other); Statens Serum Institut (Other)
Responsible Party: Sponsor-Investigator, Sabine Dieperink, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: RA-SAB2018
Record Dates: First submitted 2019-04-03; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Rheumatoid Arthritis; Staphylococcus Aureus Bacteremia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Risk Factors; Antirheumatic Agents; Biological Products; Metabolism; Adrenal Cortex Hormones; Tobacco Use Cessation Devices; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- RA patients: Incident patients with rheumatoid arthritis as identified by the Danish National Patient Registry and the rheumatology registry, DANBIO.
  Interventions: Other: Risk factors in RA cohort
- General population: All other adults, as Identified by the Civil Registration System. Patients who develop RA contribute person-years in the general population cohort until RA diagnosis
  Interventions: Other: Risk factors in general population

INTERVENTIONS:
Other: Risk factors in RA cohort
  Other Names: DMARDs (biologic and synthetic); Corticosteroids; RA disease activity; RA disease duration; Tobacco use; Joint erosions; Prosthetic joints; Other comorbid conditions and surgical/dialysis procedures
  Groups: RA patients
Other: Risk factors in general population
  Other Names: Prosthetic joints; Other comorbid conditions and surgical/dialysis procedures
  Groups: General population

SUMMARY:
Study of incidence and risk factors of staphylococcus aureus bacteremia in patients with rheumatoid arthritis compared with the general population in a nationwide cohort of all adult members of the population from 1996 until 2017 using national registries

ELIGIBILITY:
Inclusion Criteria:

* All members of the adult Danish population

Exclusion Criteria:

* Staphylococcus aureus bacteremia prior to inclusion.
* Rheumatoid arthritis diagnosed prior to inclusion.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All individuals alive and living in Denmark on December 31, 1996 as identified by the Civil Registration System are included. Individuals are dynamically included during the study period if they immigrate or turn 18. Individuals are followed up until first-time SAB, death, emigration or December 31, 2017, whichever comes first.
Sampling Method: Probability Sample
Enrollment: 6000000 (Estimated)
Dates: Start 1996-12-31 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of staphylococcus aureus bacteremia | 0-21 years
Incidence rate ratios | 0-21 years
  Comparing rheumatoid arthritis patients with the general population

SECONDARY OUTCOMES:
Risk factors of staphylococcus aureus bacteremia | 0-21 years
  Identification of risk factors both universal to both the general population and rheumatoid arthritis (RA) cohorts and RA disease specific factors (disease duration, disease activity, smoking, joint erosions, etc.)

REFERENCES:
- [Derived] Dieperink SS, Glintborg B, Oestergaard LB, Norgaard M, Benfield T, Mehnert F, Petersen A, Hetland ML. Risk factors for Staphylococcus aureus bacteremia in patients with rheumatoid arthritis and incidence compared with the general population: protocol for a Danish nationwide observational cohort study. BMJ Open. 2019 Sep 3;9(9):e030999. doi: 10.1136/bmjopen-2019-030999. PMID 31481566